CLINICAL TRIAL: NCT04258579
Title: EM/PROTECT-Hybrid: Improving Depression in Elder Mistreatment Victims
Brief Title: Trial to Test Effectiveness of Depression Intervention for Mistreated Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-09020854; P50MH113838-03 (NIH)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Results first posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Depression; Depression in Old Age; Elder Abuse; Anxiety
Keywords: Mental Health
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The investigators will be comparing data collected from this project to previously collected data from the first phase of this project, in which PROTECT was delivered only in-person.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video PROTECT (Experimental): Participants will receive PROTECT therapy once a week for 9 weeks.
  Interventions: Behavioral: PROTECT with Technology Augmentation

INTERVENTIONS:
Behavioral: PROTECT with Technology Augmentation — PROTECT is a therapeutic intervention focused on treating victims of elder abuse who are experiencing depression. PROTECT therapy will be delivered through video. Participants will be provided with a mobile device (iPhone), and a wearable device (smart watch) that will track sleep, mood, steps, and heart rate.

SUMMARY:
The investigators developed EM/PROTECT, a behavioral intervention for depressed EM (elderly mistreatment) victims, to work in synergy with EM mistreatment resolution services that provide safety planning, support services, and links to legal services. PROTECT is built on a model which postulates that chronic stress promotes dysfunction of the cognitive control (CCN) and reward networks, impairing the victims' ability to flexibly respond to the environment and limits their reward activities. PROTECT therapists work with victims to develop action plans to reduce stress, and to increase rewarding experiences. EM/PROTECT has been designed in an iterative process with community EM providers of the New York City (NYC) Department for the Aging (DFTA) to use agencies' routine PHQ-9 depression screening and referral for service. In the current study, the investigators will compare the effectiveness of EM/PROTECT with EM enriched with staff training in linking EM victims to community mental health services (EM/MH). The investigators intend to enroll 50 subjects that will participate in the study for approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* Capacity to consent (per Elder Mistreatment staff)
* Significant depression (per Elder Mistreatment staff) as indicated by a score of 10 or above on the Patient Health Questionnaire-9 (PHQ-9), a widely used screening tool routinely administered in Elder Mistreatment (EM) agency settings (the PHQ-9 has a sensitivity of 88% and a specificity of 88% for major depression)
* Need for EM services

Exclusion Criteria:

* Active suicidal ideation (Montgomery Asberg Depression Rating Scale item 10>4)
* Inability to speak English or Spanish
* Axis 1 Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) diagnoses other than unipolar depression or generalized anxiety disorder (by Structured Clinical Interview for DSM-5)
* Severe or life-threatening medical illness
* EM emergency and or referral out of EM agency (per EM staff)

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jo Anne Sirey, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this study is submitted to the National Database for Clinical Trials related to Mental Illness (NDCT). The NDCT is run by the National Institute of Health (NIH) and allows researchers studying mental health to collect and share information with each other. Researchers must apply to NIH in order to be allowed access to the data for 1 year's time; after which they must re-apply.
Time Frame: Data will be available as per the National Institute of Mental Health (NIMH) data sharing policy.
Access Criteria: Access criteria is determined by NIMH and can be requested by applying online.
URL: https://nda.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Video PROTECT
Started | 40
Completed | 27
Not Completed | 13
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Video PROTECT
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.50 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 14
  More than one race | 2
  Unknown or Not Reported | 1
Clinically Significant Depressive Symptoms, as Measured by the MADRS [Mean (Standard Deviation); unit: units on a scale] — Montgomery Asberg Depression Rating Scale. Scores on this scale range from 0 to 60, with higher scores indicating more severe depression and lower scores indicating milder depression.
  units on a scale | 23.00 (8.22)
Assessment of Quality of Life, as Measured by the WHO-QOL [Mean (Standard Deviation); unit: units on a scale] — World Health Organization-Quality Of Life scale. The overall scores range between 26-130. In all domains, higher scores indicate better health. Domain 1 measures physical health (scores range from 7-35). Domain 2 measures psychological health (scores range from 6-30). Domain 3 measures social health (scores range from 3-15). Domain 4 measures environmental health (scores range from 8-40).
  units on a scale
    Domain 1 | 21.38 (6.34)
    Domain 2 | 18.08 (5.04)
    Domain 3 | 8.45 (3.03)
    Domain 4 | 25.30 (6.26)
Assessment of Stress, as Measured by the PSS [Mean (Standard Deviation); unit: units on a scale] — Perceived Stress Scale: Overall scores range from 0-40 with higher scores indicating a more perceived stress and lower scores indicating less perceived stress.
  units on a scale | 22.45 (7.74)
Assessment of Meaningful Activities, as Measured by the BADS [Mean (Standard Deviation); unit: units on a scale] — Behavioral Activation for Depression Scale: For all domains, high scores indicate an increase of the factor or symptom described in the domain title (e.g. higher activation score means more activation). Domain 1 measures activation (scores range from 0-42). Domain 2 measures avoidance/rumination (scores range from 0-48). Domain 3 measures work and school impairment (scores range from 0-30). Domain 4 measures social impairment (scores range from 0-30).
  units on a scale
    Domain 1 | 19.89 (8.29)
    Domain 2 | 22.46 (8.57)
    Domain 3 | 16.00 (7.14)
    Domain 4 | 17.79 (7.66)

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinically Significant Depressive Symptoms as Measured by the MADRS
Description: In all conditions, the change in clinically significant depressive symptoms as measured on the Montgomery Asberg Depression Rating Scale (MADRS). Scores are categorized as following: 0 to 6 - Normal /symptom absent. 7 to 19 - Mild depression. 20 to 34 - Moderate depression. >34 - Severe depression. The scores presented for each time point are absolute values.
Time Frame: 6 weeks, 9 weeks, 12 weeks
Population: The overall number of participants analyzed was 40 at baseline, 30 at week 6, 30 at week 9, and 26 at week 12. The decline in participants analyzed at each time point is due to participant withdrawal by the study team or by their request.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Video PROTECT
Number analyzed (Participants) | 30
units on a scale
  Week 6 Outcomes | 19.13 (9.47)
  Week 9 Outcomes | 16.87 (11.69)
  Week 12 Outcomes: number analyzed (Participants) | 26
  Week 12 Outcomes | 15.00 (9.32)
Statistical Analysis 1: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 6 weeks = 19.13, 95% CI 2-sided [15.59 to 22.67]
Statistical Analysis 2: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 9 weeks = 16.87, 95% CI 2-sided [12.50 to 21.24]
Statistical Analysis 3: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 12 weeks = 15.00, 95% CI 2-sided [11.24 to 18.76]

2. Primary Outcome: Change in Assessment of Quality of Life, as Measured by the WHO-QOL
Description: In all conditions, changes in assessment of quality of life measured by the World Health Organization Quality of Life (WHO-QOL) scale. World Health Organization-Quality Of Life scale. The overall scores range between 26-130. In all domains, higher scores indicate better health. Domain 1 measures physical health (scores range from 7-35). Domain 2 measures psychological health (scores range from 6-30). Domain 3 measures social health (scores range from 3-15). Domain 4 measures environmental health (scores range from 8-40). The scores presented for each time point are absolute values.
Time Frame: 6 weeks, 9 weeks, 12 weeks
Population: The overall number of participants analyzed was 30 at week 6, 30 at week 9, and 26 at week 12. The decline in participants analyzed at each time point is due to participant withdrawal by the study team or by their request.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Video PROTECT
Number analyzed (Participants) | 30
units on a scale
  Week 6 Outcomes- Domain 1 | 22.10 (6.39)
  Week 6 Outcomes- Domain 2 | 19.90 (4.99)
  Week 6 Outcomes- Domain 3 | 8.93 (3.36)
  Week 6 Outcomes- Domain 4 | 26.63 (6.18)
  Week 9 Outcomes- Domain 1 | 22.53 (7.24)
  Week 9 Outcomes- Domain 2 | 21.00 (5.71)
  Week 9 Outcomes- Domain 3 | 8.69 (3.49)
  Week 9 Outcomes- Domain 4 | 27.38 (6.18)
  Week 12 Outcomes- Domain 1: number analyzed (Participants) | 26
  Week 12 Outcomes- Domain 1 | 22.62 (6.04)
  Week 12 Outcomes- Domain 2: number analyzed (Participants) | 26
  Week 12 Outcomes- Domain 2 | 21.58 (4.31)
  Week 12 Outcomes- Domain 3: number analyzed (Participants) | 26
  Week 12 Outcomes- Domain 3 | 9.19 (3.14)
  Week 12 Outcomes- Domain 4: number analyzed (Participants) | 26
  Week 12 Outcomes- Domain 4 | 27.81 (5.64)
Statistical Analysis 1: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 6 weeks, Domain 1 = 22.10, 95% CI 2-sided [19.70 to 24.50]
Statistical Analysis 2: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 6 weeks, Domain 2 = 19.90, 95% CI 2-sided [18.00 to 21.80]
Statistical Analysis 3: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 6 weeks, Domain 3 = 8.93, 95% CI 2-sided [7.68 to 10.18]
Statistical Analysis 4: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 6 weeks, Domain 4 = 26.63, 95% CI 2-sided [24.32 to 28.94]
Statistical Analysis 5: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 9 weeks, Domain 1 = 22.53, 95% CI 2-sided [19.87 to 25.23]
Statistical Analysis 6: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 9 weeks, Domain 2 = 21.00, 95% CI 2-sided [18.87 to 23.13]
Statistical Analysis 7: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 9 weeks, Domain 3 = 8.69, 95% CI 2-sided [7.39 to 9.99]
Statistical Analysis 8: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 9 weeks, Domain 4 = 27.38, 95% CI 2-sided [25.07 to 29.69]
Statistical Analysis 9: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 12 weeks, Domain 1 = 22.62, 95% CI 2-sided [20.18 to 25.06]
Statistical Analysis 10: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 12 weeks, Domain 2 = 21.58, 95% CI 2-sided [19.84 to 23.32]
Statistical Analysis 11: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 12 weeks, Domain 3 = 9.19, 95% CI 2-sided [7.92 to 10.46]
Statistical Analysis 12: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 12 weeks, Domain 4 = 27.81, 95% CI 2-sided [25.53 to 30.09]

3. Primary Outcome: Change in Assessment of Stress, as Measured by the PSS
Description: In all conditions, changes in assessment of stress measured by the Perceived Stress Scale (PSS) scale. Scores range from 0-40. Scores ranging from 0-13 are considered low stress, scores ranging from 14-26 are considered moderate stress, and scores ranging from 27-40 are considered high perceived stress.
Time Frame: Baseline, 6 weeks
Population: Due to participant withdrawal and loss to follow-up, the total number of participants at Week 6 was 30.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Video PROTECT
Number analyzed (Participants) | 30
units on a scale
  Baseline | 22.45 (7.74)
  Week 6 | 20.53 (7.71)
Statistical Analysis 1: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at baseline = 22.45, 95% CI 2-sided [19.56 to 25.34]
Statistical Analysis 2: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 6 weeks = 20.53, 95% CI 2-sided [17.65 to 23.41]

4. Secondary Outcome: Change in Assessment of Exposure to Meaningful Activities, as Measured by the BADS
Description: In all conditions, changes in assessment of meaningful activities measured by the Behavioral Activation for Depression Scale (BADS). Scores are divided across 4 domains: Activation subscale scores range from 0-42, Avoidance/Rumination subscale scores range from 0-48, Work/School Impairment subscale scores range from 0-30, Social Impairment subscale scores range from 0-30. For all subscales, high scores are consistent with the subscale title (e.g., high scores on Activation subscale = more activation).
Time Frame: Baseline, 6 weeks
Population: 40 subjects were analyzed at baseline. Due to participant withdrawal and loss to follow-up, the total number of participants at Week 6 was 30.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Video PROTECT
Number analyzed (Participants) | 40
units on a scale
  Baseline- Domain 1 | 19.89 (8.29)
  Baseline- Domain 2 | 22.46 (8.57)
  Baseline- Domain 3 | 16.00 (7.14)
  Baseline- Domain 4 | 17.79 (7.66)
  Week 6- Domain 1: number analyzed (Participants) | 30
  Week 6- Domain 1 | 22.79 (10.02)
  Week 6- Domain 2: number analyzed (Participants) | 30
  Week 6- Domain 2 | 26.70 (10.02)
  Week 6- Domain 3: number analyzed (Participants) | 30
  Week 6- Domain 3 | 17.45 (7.70)
  Week 6- Domain 4: number analyzed (Participants) | 30
  Week 6- Domain 4 | 20.69 (6.59)
Statistical Analysis 1: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at baseline, Domain 1 = 19.89, 95% CI 2-sided [17.24 to 22.54]
Statistical Analysis 2: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at baseline, Domain 2 = 22.46, 95% CI 2-sided [19.72 to 25.20]
Statistical Analysis 3: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at baseline, Domain 3 = 16.00, 95% CI 2-sided [13.72 to 18.28]
Statistical Analysis 4: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at baseline, Domain 4 = 17.79, 95% CI 2-sided [15.34 to 20.24]
Statistical Analysis 5: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 6 weeks, Domain 1 = 22.79, 95% CI 2-sided [19.05 to 26.53]
Statistical Analysis 6: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 6 weeks, Domain 2 = 26.70, 95% CI 2-sided [22.96 to 30.44]
Statistical Analysis 7: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 6 weeks, Domain 3 = 17.45, 95% CI 2-sided [14.57 to 20.33]
Statistical Analysis 8: Comparison: Video PROTECT; Test type: Other — Estimation only; Mean value at 6 weeks, Domain 4 = 20.69, 95% CI 2-sided [18.23 to 23.15]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Video PROTECT
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 2/40
Other Adverse Events (participants affected / at risk) | 4/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Video PROTECT (N=40)
Psychiatric Hospitalization (Psychiatric disorders) | 1 (1) — Participant was hospitalized due to a pre-existing condition.
Hospitalization due to Seizures (Nervous system disorders) | 1 (1) — Participant was hospitalized due to seizures related to a pre-existing condition.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Video PROTECT (N=40)
Emergency Room Visit (Injury, poisoning and procedural complications) | 1 (1) — Emergency room visit to assess pain from previous car accident.
Skin Irritation (Skin and subcutaneous tissue disorders) | 3 (3) — Minor skin irritation due to watch given as part of study participation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT04258579/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/79/NCT04258579/ICF_000.pdf